CLINICAL TRIAL: NCT04416243
Title: A Single-group, Feasibility, and Initial Efficacy Study of a High-intensity Interval Training Program Using Adaptive Equipment in Persons With Multiple Sclerosis Who Have Walking Disability
Brief Title: Feasibility of a High-intensity Interval Training Program in Persons With Multiple Sclerosis Who Have Walking Disability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Texas, Denton, TX (Other)
Collaborators: University of Alabama at Birmingham (Other); Berry College (Other)
Responsible Party: Principal Investigator, Stephanie Silveira, Assistant Professor, University of North Texas, Denton, TX
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018-19-24
Record Dates: First submitted 2020-05-28; First posted 2020-06-04 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; adaptive equipment; rehabilitation; recumbent stepping; high-intensity interval training
MeSH Terms: conditions — Multiple Sclerosis | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Recumbent Stepping, High-Intensity Interval Training (Experimental)
  Interventions: Behavioral: Recumbent Stepping, High-Intensity Interval Training

INTERVENTIONS:
Behavioral: Recumbent Stepping, High-Intensity Interval Training — The intervention will involve 12 weeks of supervised, progressive (i.e., intensity increases after midpoint testing based on reassessment of aerobic fitness) HIIT sessions two to three times per week. HIIT exercise sessions will be manualized and led by exercise leaders. Secondary outcomes testing will occur at baseline (week 0), midpoint (following week 6 of training), and post-intervention (following week 12 of training).
  The individual HIIT sessions will involve 10 cycles of 60s intervals at the wattage associated with 90% VO2peak followed by 60s of active recovery intervals at 15 watts, totaling 20 min in length. All exercise sessions will begin and end with a 5-minute warm-up and cool-down, respectively. Required power output for each interval of the exercise session will be individualized and completely automated. VO2peak from baseline and midpoint testing will be used to determine exercise intensity for weeks 1-6 and weeks 7-12, respectively.

SUMMARY:
There is considerable evidence to support the efficacy of moderate intensity continuous (MIC) exercise benefitting clinically-relevant outcomes in persons with multiple sclerosis (MS). However, persons with MS who have walking impairments (pwMS-wd) are severely deconditioned and may achieve superior benefits by engaging in high-intensity interval training (HIIT), especially while utilizing adaptive equipment, such as with recumbent arm/leg stepping (RSTEP). Of the published studies on HIIT in MS, HIIT yielded significant improvements in cardiorespiratory fitness in all but one study. In those studies that directly compared HIIT to MIC exercise, the data indicated a potential superiority of HIIT as compared to MIC in improving physiological conditioning in a time efficient manner. However, this evidence is specific to those with MS with mild to moderate disability engaging in cycle/arm ergometry and an investigation of HIIT in pwMS-wd is needed as the feasibility and potential benefits of engaging in HIIT in pwMS-wd is relatively unknown.

The primary aim of the proposed study is to assess the feasibility of a 12-week, RSTEP HIIT program in pwMS-wd. The secondary aim is to examine changes in aerobic fitness, physical activity, ambulation, upper arm function, cognition, fatigue, and depressive symptoms as clinically-relevant efficacy outcomes following the 12-week, RSTEP HIIT intervention. It is hypothesized that the intervention will be feasible and lead to positive changes in aerobic fitness, physical activity, ambulation, upper arm function, cognition, fatigue, and depressive symptoms. This work is informed by recently published data, which indicate that a single bout of RSTEP HIIT taxes the cardiorespiratory system significantly more than MIC exercise, yet without untoward effects on walking, gait, cognition, mood, or enjoyment. These data suggest that RSTEP HIIT may be an acceptable, safe, and tolerable stimulus for chronic exercise training.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or over
* a self-reported diagnosis of multiple sclerosis
* self-reported Expanded Disability Status Scale (EDSS) score < 8.0 or Patient Determined Disability Steps (PDDS) scale score ≤ 7.0
* relapse free in past 30 days
* willing and able to visit Berry College or University of North Texas on three testing occasions and twenty four training occasions
* asymptomatic status for maximal exercise testing; (g) physician approval for undertaking exercise testing
* a self-reported ability to speak, read, and understand English

Exclusion Criteria:

* Any persons who do not meet the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-12-19 (Actual); Primary Completion 2022-12-14 (Actual); Study Completion 2022-12-14 (Actual)

PRIMARY OUTCOMES:
Recruitment, Retention, and Adherence Rates | From recruitment to end of treatment at 12 weeks.
  Participant recruitment, retention, and adherence rates will be recorded.
Time Needs | From recruitment to end of treatment at 12 weeks.
  Staff training, communication, recruitment, and intervention time will be recorded.
Monetary Needs | From recruitment to end of treatment at 12 weeks.
  Monetary research costs will be recorded.
Data Management and Safety Reporting | From recruitment to end of treatment at 12 weeks.
  Time from submission of Institutional Review Board application to approval will be recorded. All time spent collecting, entering, and checking data will be recorded.
Participant Burden Reporting | From recruitment to end of treatment at 12 weeks.
  Participants' experience, burden, and perceptions will be assessed via a short survey at the end of the 12 weeks.
Safety Reporting | From recruitment to end of treatment at 12 weeks.
  Adverse events, serious adverse events, and clinical emergencies will be recorded.

SECONDARY OUTCOMES:
Change in Aerobic Capacity | Week 0, Following Week 6, Following Week 12
  Participants will complete a standardized graded maximal exercise step on a recumbent stepper. The highest recorded 30-second volume of oxygen consumption (VO2) value will be recorded as VO2peak, expressed in mL/kg/min, when at least 1 of the following criteria are satisfied: (1) respiratory exchange ratio 1.10 or greater; (2) peak heart rate within 10 beats per minute of age-predicted maximum(i.e., 220-age); or (3) ratings of perceived exertion of 7 or greater.
Change in 6-Minute Walk Distance | Week 0, Following Week 6, Following Week 12
  Participants will walk for a total of 6 minutes along a single course 75-feet in length with two, 180-degree turns. Total distance travelled (ft) will be recorded.
Change in 25-Foot Walk Speed | Week 0, Following Week 6, Following Week 12
  Participants will be instructed to walk as fast as possible along a 25-foot path. Participants time recorded as walking speed (ft/s) will be collected twice. The average of the two trials will be reported.
Change in Sedentary, Light, and Moderate-to-Vigorous Counts of Physical Activity | Week 0, Following Week 6, Following Week 12
  Participants will be asked to wear an accelerometer for 7 consecutive days for a minimum of 10 hours of wear time. Using the accelerometer software, sedentary, light, and moderate-to-vigorous counts of physical activity will be generated based on disability status.
Change in the Brief International Cognitive Assessment in MS Scores | Week 0, Following Week 6, Following Week 12
  Participants will complete the oral version of the Symbol Digit Modalities Test, the first five recall trials of the California Verbal Learning Test-2, and the first three recall trials of the Brief Visuospatial Memory Test-Revised. The Symbol Digit Modalities Test reports the correct number of responses with a maximum score of 110. The California Verbal Learning test reports the total number of correct words identified over five trials, with a maximum score of 90. The Brief Visuospatial Memory Test-Revised reports the total raw score across the three trials, with a maximum score of 36.
Change in 9-Hole Peg Test Score | Week 0, Following Week 6, Following Week 12
  Participants are instructed to pick up pegs and place them one at a time into one of nine holes as fast as possible and then to remove the pegs, one at a time, with the same hand. The time (s) to complete this activity will be recorded and averaged on two trials for the dominant hand and then the non-dominant hand.
Change in Fatigue Scores | Week 0, Following Week 6, Following Week 12
  Participants will be asked to complete the Fatigue Severity Scale, which is a self-report measure comprised of 9 items that assess the severity of fatigue symptoms. This Likert scale ranges from 1 (strongly disagree) and 7 (strongly agree) and measures the degree of fatigue severity over the past week. All items will be summed for a final score with higher scores indicating greater fatigue severity and a maximum score of 63.
Change in Depressive Symptoms Scores | Week 0, Following Week 6, Following Week 12
  Depressive symptoms will be measured by the Depression sub-scale of the Hospital Anxiety and Depression Scale (HADS-D). The HADS-D includes 7 items that measure depression and are rated on a 4-point scale ranging between 0 (not at all) to 3 (most of the time). Positively worded items are reverse-scored and then added with negatively worded items to create a total sum with a maximum value of 21.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie L Silveira, PhD, Principal Investigator — University of North Texas Health Science Center
Locations (1):
- University of North Texas, Denton, Texas, United States

REFERENCES:
- [Derived] Hubbard EA, Motl RW, Elmer DJ. Feasibility and initial efficacy of a high-intensity interval training program using adaptive equipment in persons with multiple sclerosis who have walking disability: study protocol for a single-group, feasibility trial. Trials. 2020 Nov 25;21(1):972. doi: 10.1186/s13063-020-04887-x. PMID 33239079